CLINICAL TRIAL: NCT01905163
Title: Prospective Study Assessing the Feasibility of Interval Debulking Surgery by Laparoscopy for Peritoneal Carcinomatosis of Ovarian Origin, Tubal or Primary Peritoneal, in Chemosensitive Patients Treated by Neoadjuvant Chemotherapy.
Brief Title: Feasibility of Interval Debulking Surgery by Laparoscopy for Peritoneal Carcinosis in Chemosensitive Patients
Acronym: CILOVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-A01391-42
Record Dates: First submitted 2013-07-09; First posted 2013-07-23 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cavity Cancer
Keywords: Laparoscopy, interval debulking surgery
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- laparoscopic management (Experimental): Tumor Debulking Surgery by laparoscopy
  Interventions: Procedure: Tumor Debulking Surgery by laparoscopy

INTERVENTIONS:
Procedure: Tumor Debulking Surgery by laparoscopy

SUMMARY:
This prospective nonrandomized multicenter phase II study, will evaluate the possibility of performing a laparoscopic interval debulking after a minimum of 3 cycles of chemotherapy in highly chemo-sensitive patients with advanced ovarian, tubal cancer or primary peritoneal.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years
* performance status WHO < 2
* Epithelial ovarian, fallopian tubes or primary peritoneal carcinoma (histologically confirmed)
* Unresectable disease because of FIGO stage IV disease proven by imaging (CT Scan or PET CT) and/or diffuse extensive carcinosis considered unresectable for advanced FIGO stage IIIc; or patients unable to support a radical primary surgery because of age, comorbidities or altered general condition.
* No previous debulking surgery before neoadjuvant chemotherapy.
* Patients treated with a minimum of 3 cycles of platinum-based neoadjuvant chemotherapy.
* Response to chemotherapy was radiologically confirmed (Scan-TAP) prior to interval surgery:

No evidence of peritoneal supra-mesocolic carcinomatosis ; Residual pelvic masses smaller than 10 cm ; Absence of suspect supra-centimeter retroperitoneal lymphadenopathy

* able to read, write and understand French.
* Member of a Social Security scheme.
* written informed consent.

Exclusion Criteria:

* Patient unable to support laparoscopy
* psychiatric condition or social or geographic situation that would impede appropriate study participation
* Concomitant participation in another clinical trial evaluating surgical treatment (interfering with the evaluation of the main endpoint)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-08; Primary Completion 2016-08 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
the rate of conversion to laparotomy | surgery
  Feasibility of the surgical laparoscopic management of interval debulking surgery will be assessed by the rate of conversion to laparotomy.

SECONDARY OUTCOMES:
Port site metastases | during 1 year post surgery
Morbidity: intraoperative and postoperative complications | during surgery and 1 year post surgery
Pain | during the hospital stay (an expected average of 5 days), at 1 week, 1 month, 3 and 6 months post surgery
Quality of life using EORTC QLQ-C30 | before surgery (an expected average of 7 days before surgery), 1 week , 1 month, 3 and 6 months post-surgery
Economic evaluation | 1 year post-surgery
  economic evaluation will be assess by a quantification of the additional costs of surgery, duration and cost of hospitalization, number of possible re-interventions or hospitalizations.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe POMEL, Pr, Principal Investigator — Centre Jean Perrin
Locations (10):
- France (10):
  - Institut de Cancerologie de l'Ouest, site Paul Papin, Angers
  - CHU Estaing, Clermont-Ferrand
  - Centre Jean Perrin, Clermont-Ferrand
  - Institut Paoli Calmettes, Marseille
  - Institut Curie, Paris
  - Hôpital Européen Georges-Pompidou, Paris
  - Institut Curie - Hôpital René Huguenin, Saint-Cloud
  - Institut de Cancérologie de L'Ouest, Saint-Herblain
  - Hôpital de Hautepierre, Strasbourg
  - Institut Claudius Regaud, Toulouse